CLINICAL TRIAL: NCT00798434
Title: A 24-Week, Multi-Centre Trial, Comprising A 12-Week, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Phase Followed By A 12-Week Open-Label Phase, To Evaluate The Efficacy And Safety Of A Fesoterodine Flexible Dose Regimen In Elderly Patients With Overactive Bladder.
Brief Title: A Study to Compare the Effectiveness and Safety of Fesoterodine and Placebo in an Elderly Population of Patients Who go to the Toilet Very Frequently Due to Overactive Bladder.
Acronym: SOFIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0221045
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-11

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder syndrome; fesoterodine; elderly; flexible dose regimen; urgency; frequency; urge urinary incontinence; anticholinergic; antimuscarinic
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Active Comparator): Flexible dose regimen of placebo once daily. The dose can be increased after 4 weeks if clinically indicated. Subsequently the dose can be reduced to the original dose if clinically indicated.
  Interventions: Drug: Placebo
- Fesoterodine (Active Comparator): Flexible dose regimen of fesoterodine fumarate 4mg once daily. The dose can be increased to 8mg once daily after 4 weeks if clinically indicated. Subsequently the dose can be reduced to 4mg if clinically indicated.
  Interventions: Drug: Fesoterodine fumarate

INTERVENTIONS:
Drug: Placebo — placebo administered orally in the morning or evening.
  Arms: Placebo
Drug: Fesoterodine fumarate — Fesoterodine fumarate is an antimuscarinic drug recently approved by the European Medicines Evaluation Agency for treatment of symptoms of overactive bladder syndrome.
  Other Names: Toviaz
  Arms: Fesoterodine

SUMMARY:
The drug being studied, fesoterodine fumarate helps prevent the bladder neck opening at unwanted times and has been shown to help patients with overactive bladder syndrome pass urine less frequently than before treatment. It is postulated that this drug will also prove effective in elderly patients (aged > 65 years) and that the ability to change dose between 4 and 8mg will allow each patient to have an optimised treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥65 years old.
* Overactive bladder symptoms for at least 3 months prior to study start.
* Eight or more micturitions per 24 hours as confirmed by diary records

Exclusion Criteria:

* Predominant Stress Urinary Incontinence
* Active or recurrent bladder infections
* Other bladder and genital conditions that could be the predominant cause of symptoms or interfere with treatment assessment and success.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 794 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- Pfizer Investigational Site, Vienna, Austria
- Belgium (4):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Kortrijk
- Denmark (2):
  - Pfizer Investigational Site, Aarhus N
  - Pfizer Investigational Site, Glostrup Municipality
- Finland (5):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kouvola
  - Pfizer Investigational Site, OYS
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, München
- Israel (2):
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Jerusalem
- Italy (2):
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Terracina, LT
- Norway (4):
  - Pfizer Investigational Site, Hamar
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Trondheim
  - Pfizer Investigational Site, Tønsberg
- Portugal (3):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Galanta
  - Pfizer Investigational Site, Kosice - Saca
  - Pfizer Investigational Site, Košice
- Spain (5):
  - Pfizer Investigational Site, Martorell, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Getafe, Madrid
  - Pfizer Investigational Site, Manacor, Palma de Mallorca
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (5):
  - Pfizer Investigational Site, Eslöv
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Norrköping
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site, Frauenfeld, Switzerland
- Turkey (Türkiye) (4):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
  - Pfizer Investigational Site, Samsun
- United Kingdom (6):
  - Pfizer Investigational Site, Bexhill-on-Sea, East Sussex
  - Pfizer Investigational Site, Leytonstone, London
  - Pfizer Investigational Site, Harrow, Middlesex
  - Pfizer Investigational Site, High Heaton, Newcastle upon Tyne
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, London

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Wagg A, Khullar V, Michel MC, Oelke M, Darekar A, Bitoun CE. Long-term safety, tolerability and efficacy of flexible-dose fesoterodine in elderly patients with overactive bladder: open-label extension of the SOFIA trial. Neurourol Urodyn. 2014 Jan;33(1):106-14. doi: 10.1002/nau.22383. Epub 2013 Mar 4. PMID 23460503
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221045&StudyName=A%20study%20to%20compare%20the%20effectiveness%20and%20safety%20of%20fesoterodine%20and%20placebo%20in%20an%20elderly%20population%20of%20patients%20who%20go%20to%20the%20toi

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Fesoterodine: Participants received 12 weeks of matched placebo (double-blinded), followed by 12 weeks of fesoterodine 4 milligrams (mg) once daily (open-label). During study, participants permitted 1 dose increase to fesoterodine 8 mg daily (and 1 decrease from 8 mg back to 4 mg, if necessary).
- Fesoterodine/Fesoterodine: Participants received 12 weeks of fesoterodine 4 mg once daily (double-blinded), followed by 12 weeks of fesoterodine 4 mg once daily (open-label). During study, participants permitted 1 dose increase to fesoterodine 8 mg daily (and 1 decrease from 8 mg back to 4 mg, if necessary).
Period: Double-Blind
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Started | 396 | 398
Received Treatment | 393 | 392
Completed | 341 | 314
Not Completed | 55 | 84
Not completed — Adverse Event | 22 | 46
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 8 | 12
Not completed — Withdrawal by Subject | 17 | 14
Not completed — Protocol Violation | 1 | 4
Not completed — Did Not Meet Entrance Criteria | 2 | 1
Not completed — Other | 1 | 0
Not completed — Not Treated | 3 | 6
Period: Open-Label
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Started | 341 | 314
Received Treatment | 341 | 313
Completed | 299 | 282
Not Completed | 42 | 32
Not completed — Adverse Event | 33 | 11
Not completed — Lack of Efficacy | 5 | 11
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 1 | 2
Not completed — Not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Fesoterodine: Participants received 12 weeks of matched placebo (double-blinded), followed by 12 weeks of fesoterodine 4 mg once daily (open-label). During study, participants permitted 1 dose increase to fesoterodine 8 mg daily (and 1 decrease from 8 mg back to 4 mg, if necessary).
- Total: Total of all reporting groups
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine | Total
Number analyzed (Participants) | 393 | 392 | 785
Age, Customized [Number; unit: participants]
  65-75 years | 267 | 264 | 531
  76-84 years | 114 | 116 | 230
  greater than or equal to 85 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 213 | 418
  Male | 188 | 179 | 367
Patient Perception of Bladder Condition (PPBC) at Baseline [Number; unit: Participants] — Participants who contributed to baseline score; PPBC: self-administered, single-item, questionnaire asked participants to describe their perception of their bladder-related problems; Rated on a 6-point scale: 1=no problems at all, 2=some very minor problems, 3=some minor problems, 4=moderate problems, 5=severe problems, 6=many severe problems
  Participants
    no problems at all | 0 | 0 | 0
    some very minor problems | 1 | 0 | 1
    some minor problems | 2 | 2 | 4
    some moderate problems | 185 | 190 | 375
    severe problems | 157 | 158 | 315
    many severe problems | 37 | 23 | 60
Micturition-Related Urgency Episodes per 24 Hours [Median (Full Range); unit: Episodes per 24 hours] — Micturition-related urgency episodes per 24 hours defined as those with Urinary Sensation Scale (USS) rating of >=3 marked for corresponding micturition in diary. USS rating of 3: Moderate feeling of urgency, 4: Severe feeling of urgency, 5: Unable to hold; leak urine.
  Episodes per 24 hours | 8.7 [0.0 to 28.7] | 8.5 [1.3 to 21.0] | 8.7 [0.0 to 28.7]
Severe Micturition-Related Urgency Episodes per 24 Hours [Median (Full Range); unit: Episodes per 24 hours] — Severe micturition-related urgency episodes defined as those with USS rating >=4. USS rating of 4: Severe feeling of urgency and 5: Unable to hold; leak urine.
  Episodes per 24 hours | 3.0 [0.0 to 28.7] | 2.7 [0.0 to 19.0] | 2.7 [0.0 to 28.7]
Micturitions per 24 Hours [Median (Full Range); unit: Episodes per 24 hours] — Micturitions included episodes of voluntary micturition and episodes of Urgency Urinary Incontinence (UUI).
  Episodes per 24 hours | 11.5 [7.0 to 28.7] | 11.3 [7.5 to 25.7] | 11.3 [7.0 to 28.7]
Nocturnal Micturitions per 24 Hours [Median (Full Range); unit: Episodes per 24 hours] — Nocturnal micturitions defined as micturitions with USS rating 1-5 that occurred between time participant went to bed and time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
  Episodes per 24 hours | 2.7 [0.0 to 10.0] | 2.7 [0.0 to 12.3] | 2.7 [0.0 to 12.3]
UUI Episodes per 24 Hours [Median (Full Range); unit: Episodes per 24 hours] — UUI episodes defined as those with the USS rating of 5 (unable to hold; leak urine) in the diary.
  Episodes per 24 hours | 0.0 [0.0 to 26.7] | 0.0 [0.0 to 14.3] | 0.0 [0.0 to 26.7]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Micturition-Related Urgency Episodes Per 24 Hours at Week 12
Description: Number of micturition-related urgency episodes per 24 hours calculated as number of micturitions with USS rating of greater than or equal to (>=) 3 divided by number of days that diary data was collected at that visit. USS ranged 1 to 5 (1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine). Change = observation minus baseline, where lower scores were an improvement/decrease in micturition-related urgency episodes.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS)=randomized participants who took at least 1 dose of double-blind (DB) treatment, had baseline and post-baseline efficacy data for at least 1 endpoint and at least 1 time point during DB treatment; number of participants analyzed (n)=participants with evaluable data at the specified time point.
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours
Groups:
- Placebo: Participants received matched placebo once daily from baseline to Week 12 (double-blinded) with 1 permitted sham dose increase (and 1 sham decrease if necessary).
- Fesoterodine: Participants received fesoterodine 4 mg once daily from baseline to Week 12 (double-blinded) with 1 permitted dose increase to fesoterodine 8 mg daily (and 1 decrease from 8 mg back to 4 mg, if necessary).
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 381 | 374
Episodes per 24 hours
  Baseline (n=381, 374) | 8.80 (3.97) | 8.48 (3.62)
  Change at Week 12 (n=356, 338) | -2.48 (4.53) | -3.84 (4.10)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Based on a 2-sided t-test (5% significance). Null hypothesis: no difference in mean change in mean micturition-related urgency episodes per 24 hours at Week 12 for the 2 groups. Last observation carried forward (LOCF) method used for statistical analyses of the FAS (change from baseline to Week 12); Test type: Superiority or Other; p < 0.0001, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline urgency episodes; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-2.12 to -0.97], Standard Error of Mean 0.29

2. Secondary Outcome: Percent Change From Baseline in Micturition-Related Urgency Episodes Per 24 Hours at Weeks 4, 8, and 12
Description: Micturition-related urgency episodes per 24 hours defined as those with USS Scale rating of >=3 marked for corresponding micturition in diary. USS rating of 3: Moderate feeling of urgency, 4: Severe feeling of urgency, 5: Unable to hold; leak urine. Percent change calculated as: 100* (Urgency Episode at Week x - baseline)/baseline. Change = observation minus baseline, where lower scores were an improvement/decrease in micturition-related urgency episodes.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: FAS;N=participants with evaluable data; n=participants with evaluable data at specific time point. LOCF method used for statistical analyses of the FAS (change from baseline to Week 12).
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Percent change
  Change at Week 4 (n=365, 356) | 6.7 [0.0 to 29.0] | 5.3 [0.0 to 20.7]
  Change at Week 8 (n=349, 331) | 5.7 [0.0 to 26.0] | 4.3 [0.0 to 18.7]
  Change at Week 12 (n=356, 338) | 5.3 [0.0 to 27.3] | 3.7 [0.0 to 21.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, 2-sided Van Elteren's test; Median Difference (Final Values) = -14.44, 95% CI 2-sided [-14.67 to -14.25] — Hodges-Lehman estimate of median treatment difference and confidence interval (CI)

3. Secondary Outcome: Change From Baseline in Mean Number of Severe Micturition-Related Urgency Episodes Per 24 Hours at Weeks 4, 8, and 12
Description: Severe micturition-related urgency episodes defined as those with the USS rating >=4. USS rating of 4: Severe feeling of urgency and 5: Unable to hold; leak urine. Change = observation minus baseline, where lower scores were an improvement/decrease in severity of micturition-related urgency episodes.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: FAS; N=participants with evaluable data; n=participants with evaluable data at specific time point. LOCF method used for statistical analyses of the FAS (change from baseline to Week 12).
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 381 | 374
Episodes per 24 hours
  Baseline (n=381, 374) | 4.11 (4.24) | 3.53 (3.40)
  Change at Week 4 (n=365, 356) | -0.96 (3.39) | -1.81 (2.96)
  Change at Week 8 (n=349, 331) | -1.53 (3.79) | -2.12 (3.07)
  Change at Week 12 (n=356, 338) | -1.78 (3.85) | -2.43 (3.14)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p = 0.0001, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline severe urgency episodes; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.28 to -0.42], Standard Error of Mean 0.22

4. Secondary Outcome: Percent Change From Baseline of Severe Micturition-Related Urgency Episodes Per 24 Hours at Weeks 4, 8, and 12
Description: Severe micturition-related urgency episodes defined as those with USS rating >=4. USS rating of 4: Severe feeling of urgency and 5: Unable to hold; leak urine. Change = observation minus baseline, where lower scores were an improvement/decrease in severity of micturition-related urgency.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Percent change
  Change at Week 4 (n=365, 356) | -0.7 [-16.7 to 14.7] | -1.3 [-16.0 to 11.3]
  Change at Week 8 (n=349, 331) | -1.0 [-23.3 to 15.3] | -1.7 [-17.3 to 6.3]
  Change at Week 12 (n=356, 338) | -1.3 [-23.3 to 17.3] | -2.0 [-17.3 to 7.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p = 0.0005, 2-sided Van Elteren's test; Median Difference (Final Values) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Hodges-Lehman estimate of median treatment difference and CI

5. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Weeks 4, 8, and 12
Description: Micturitions included episodes of voluntary micturition and episodes of UUI, defined as those micturitions with USS rating of 5 (unable to hold; leak urine) in the diary of participants with UUI at baseline. Change = observation minus baseline, where lower scores were an improvement/decrease in micturitions.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: FAS; n=participants with evaluable data at specific time point. LOCF method used for statistical analyses of the FAS (change from baseline to Week 12).
Measure: Mean (Standard Deviation); unit: Micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Micturitions per 24 hours
  Baseline (n=382, 374) | 12.10 (3.12) | 11.89 (2.90)
  Change at Week 4 (n=366, 356) | -0.69 (2.26) | -1.47 (2.19)
  Change at Week 8 (n=349, 331) | -1.11 (2.37) | -1.95 (2.33)
  Change at Week 12 (n=359, 338) | -1.15 (2.56) | -2.09 (2.33)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline number of micturitions; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-1.33 to -0.64], Standard Error of Mean 0.18

6. Secondary Outcome: Percent Change From Baseline in Micturitions Per 24 Hours at Weeks 4, 8, and 12
Description: Micturitions included episodes of voluntary micturition and episodes of UUI. Change = observation minus baseline, where lower scores were an improvement/decrease in micturitions.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 5
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Percent change
  Change at Week 4 (n=366, 356) | -0.7 [-7.7 to 9.7] | -1.3 [-11.7 to 11.7]
  Change at Week 8 (n=349, 331) | -1.0 [-7.3 to 10.3] | -1.7 [-12.3 to 9.3]
  Change at Week 12 (n=359, 338) | -1.3 [-7.7 to 10.0] | -2.0 [-12.7 to 7.0]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, 2-sided Van Elteren's test; Median Difference (Final Values) = -7.31, 95% CI 2-sided [-7.40 to -7.19]

7. Secondary Outcome: Change From Baseline in Number of Nocturnal Micturitions Per 24 Hours at Weeks 4, 8, and 12
Description: Nocturnal micturitions defined as micturitions with USS rating 1-5 that occurred between time participant went to bed and time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. Calculated as number of nocturnal micturitions divided by number of diary days collected at that visit. Change = observation minus baseline, where lower scores were an improvement/decrease in nocturnal micturitions.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Micturitions per 24 hours
  Baseline (n=382, 374) | 2.92 (1.46) | 2.80 (1.47)
  Change at Week 4 (n=366, 356) | -0.22 (1.15) | -0.38 (0.99)
  Change at Week 8 (n=349, 331) | -0.30 (1.13) | -0.51 (1.03)
  Change at Week 12 (n=359, 338) | -0.33 (1.15) | -0.55 (1.13)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p = 0.0026, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline number of night-time micturitions; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.40 to -0.09], Standard Error of Mean 0.08

8. Secondary Outcome: Percent Change From Baseline in Nocturnal Micturitions Per 24 Hours at Weeks 4, 8, and 12
Description: Nocturnal micturitions defined as micturitions with USS rating 1-5 that occurred between time participant went to bed and time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. Change = observation minus baseline, where lower scores were an improvement/decrease in nocturnal micturitions.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: FAS; n=participants with evaluable data at specific time point. LOCF method was used for the statistical analyses of the FAS (change from baseline to Week 12).
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Percent change
  Change at Week 4 (n=366, 356) | -0.3 [-5.0 to 8.3] | -0.3 [-4.7 to 3.7]
  Change at Week 8 (n=349, 331) | -0.3 [-4.0 to 6.7] | -0.7 [-4.3 to 4.0]
  Change at Week 12 (n=359, 338) | -0.3 [-4.0 to 6.3] | -0.7 [-5.3 to 3.0]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p = 0.0012, 2-sided Van Elteren's test; Median Difference (Final Values) = -9.52, 95% CI 2-sided [-9.52 to -9.09]

9. Secondary Outcome: Change From Baseline in Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Weeks 4, 8, and 12
Description: UUI episodes defined as those with USS rating of 5 (unable to hold; leak urine) in the diary. Change = observation minus baseline, where lower scores were an improvement/decrease in UUI episodes.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: Episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 381 | 374
Episodes per 24 hours
  Baseline (n=381, 374) | 0.0 [0.0 to 26.7] | 0.0 [0.0 to 14.3]
  Change at Week 4 (n=365, 356) | 0.0 [-14.3 to 22.3] | 0.0 [-13.7 to 8.3]
  Change at Week 8 (n=349, 331) | 0.0 [-12.3 to 22.0] | 0.0 [-14.3 to 2.7]
  Change at Week 12 (n=356, 338) | 0.0 [-14.0 to 22.3] | 0.0 [-10.3 to 7.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p = 0.1005, Van-Elteren's Test — The protocol-defined analysis (ANOVA, parametric) not presented because normality assumptions were not met, instead an alternative analysis (Van-Elteren'ts test, non-parametric) as defined in the statistical analysis plan presented; Hodges-Lehman estimate = 0.00, 95% CI 2-sided [0.00 to 0.00] — Hodges-Lehman estimate of median treatment difference and CI

10. Secondary Outcome: Percent Change From Baseline of UUI Episodes Per 24 Hours at Weeks 4, 8, and 12
Description: UUI episodes defined as those with the USS rating of 5 (unable to hold; leak urine)in the diary. Change = observation minus baseline, where lower scores were an improvement/decrease in UUI episodes.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: FAS; N=participants with evaluable data; n=participants with evaluable data at specific time point. LOCF method was used for the statistical analyses of the FAS (change from baseline to Week 12).
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Percent change
  Change at Week 4 (n=365, 356) | 0.0 [0.0 to 22.7] | 0.0 [0.0 to 9.3]
  Change at Week 8 (n=349, 331) | 0.0 [0.0 to 23.3] | 0.0 [0.0 to 5.7]
  Change at Week 12 (n=356, 338) | 0.0 [0.0 to 22.7] | 0.0 [0.0 to 14.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p = 0.0218, 2-sided Van Elteren's test; Median Difference (Final Values) = 0.00, 95% CI 2-sided [0.00 to 0.00]

11. Secondary Outcome: Change From Baseline in Daily Sum Rating in USS at Weeks 4, 8, and 12
Description: USS total range 1 to 5 (1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine). Change = observation minus baseline, where lower scores were an improvement/decrease in urinary sensation.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 381 | 374
Scores on a scale
  Baseline (n=381, 374) | 37.55 (13.95) | 36.07 (11.16)
  Change at Week 4 (n=365, 356) | -4.35 (11.7) | -8.52 (10.0)
  Change at Week 8 (n=349, 331) | -6.53 (12.5) | -10.81 (10.7)
  Change at Week 12 (n=356, 338) | -7.33 (12.7) | -11.59 (10.7)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; Covariates were treatment, study center, dosing time, age category, and daily sum rating of USS at baseline; Mean Difference (Final Values) = -4.70, 95% CI 2-sided [-6.30 to -3.10], Standard Error of Mean 0.81

12. Secondary Outcome: Percentage of Participants Who Were Incontinent at Baseline and Became Dry
Description: Percentage of participants who had at least 1 UUI episode during baseline period and were dry (no UUI episodes) in the 3 days prior to study visits at week 8 and 12. UUI episodes defined as those with USS rating of 5 (unable to hold; leak urine) in the diary.
Time Frame: Weeks 8 to 12
Population: FAS; N=number of participants with evaluable data. LOCF method was used for the statistical analyses of the FAS (change from baseline to Week 12).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 160 | 158
Percentage of participants | 45.0 | 53.2
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; LOCF; Test type: Superiority or Other; p = 0.1113, Regression, Logistic — Logistic regression determined the odds of improvement versus no improvement in dryness, where improvement was defined as dry at both weeks 8 and 12 relative to baseline incontinence; Covariates were treatment, study center, dosing time, and age category; Odds Ratio (OR) = 1.515, 95% CI 2-sided [0.909 to 2.528]

13. Secondary Outcome: Change From Baseline in Number of Skin Protective Agents Used by Participants at Weeks 4, 8, and 12
Description: Skin protective agents included incontinence pads, barrier creams, and powders. Change = observation minus baseline, where lower scores were an improvement/decrease in protective skin agents used.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Skin protective agents
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 374 | 369
Skin protective agents
  Incontinence pads at Baseline (n=374, 369) | 1.49 (2.70) | 1.35 (2.01)
  Incontinence pads Change at Week 4 (n=360, 350) | -0.20 (1.97) | -0.27 (1.33)
  Incontinence pads Change at Week 8 (n=342, 326) | -0.15 (2.01) | -0.38 (1.57)
  Incontinence pads Change at Week 12 (n=350, 332) | -0.16 (1.98) | -0.50 (1.35)
  Creams at Baseline (n=374, 368) | 0.12 (0.72) | 0.16 (0.68)
  Creams Change at Week 4 (n=360, 349) | -0.01 (0.55) | -0.02 (0.39)
  Creams Change at Week 8 (n=342, 325) | 0.06 (0.60) | -0.03 (0.47)
  Creams Change at Week 12 (n=350, 331) | 0.04 (0.41) | -0.03 (0.54)
  Powder at Baseline (n=374, 368) | 0.03 (0.29) | 0.02 (0.23)
  Powder Change at Week 4 (n=360, 349) | 0.03 (0.27) | -0.02 (0.24)
  Powder Change at Week 8 (n=342, 325) | 0.03 (0.39) | -0.01 (0.29)
  Powder Change at Week 12 (n=350, 331) | 0.03 (0.44) | -0.02 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Incontinence pads at Week 12 LOCF; Test type: Superiority or Other; p = 0.0230, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline number of pads per 24 hours; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.47 to -0.04], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Creams at Week 12 LOCF; Test type: Superiority or Other; p = 0.0909, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline number of creams per 24 hours; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.12 to 0.01], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Powder at Week 12 LOCF; Test type: Superiority or Other; p = 0.2039, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline number of powders per 24 hours; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.08 to 0.02], Standard Error of Mean 0.03

14. Secondary Outcome: Percentage of Participants With Improvement at Week 12
Description: Patient Treatment Benefit Scale (PTBS): single-item scale assessed fesoterodine efficacy and safety in participants with overactive bladder. Participants asked to compare their present condition with their condition before start of trial: "My condition has been: 1=Greatly Improved; 2=Improved; 3=Not Changed; 4=Worsened, During Treatment." Improvement was defined as a rating of 1 or 2.
Time Frame: Week 12
Population: FAS; N=participants with evaluable data. LOCF method was used for the statistical analyses of the FAS (change from baseline to Week 12).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 340 | 334
Percentage of participants | 42.9 | 67.7
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Covariates were treatment, study center, dosing time, and age category; Odds Ratio (OR) = 3.096, 95% CI 2-sided [2.181 to 4.395]

15. Secondary Outcome: Change From Baseline in Patient Perception of Bladder Condition (PPBC) at Week 4
Description: PPBC: self-administered, single-item, questionnaire that asked participants to describe their perception of their bladder-related problems. PPBC assessment rated on a 6-point scale: 1=no problems at all, 2=some very minor problems, 3=some minor problems, 4=moderate problems, 5=severe problems, 6=many severe problems. Change = observation minus baseline. Results categorized as Deterioration (score difference ≥1), No Change (score difference=0), Improvement (score difference less than [<]0).
Time Frame: Baseline and Week 4
Population: FAS; N=participants with evaluable data
Measure: Number; unit: Participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 370 | 360
Participants
  Improvement | 168 | 192
  No Change | 202 | 168
  Deterioration | 40 | 16

16. Secondary Outcome: Change From Baseline in PPBC at Week 8
Description: PPBC: self-administered, single-item, questionnaire that asked participants to describe their perception of their bladder-related problems. PPBC assessment rated on a 6-point scale: 1=no problems at all, 2=some very minor problems, 3=some minor problems, 4=moderate problems, 5=severe problems, 6=many severe problems. Change = observation minus baseline. Results categorized as Deterioration (score difference ≥1), No Change (score difference=0), Improvement (score difference <0).
Time Frame: Baseline and Week 8
Population: FAS; N=participants with evaluable data
Measure: Number; unit: Participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 351 | 329
Participants
  Improvement | 185 | 210
  No Change | 166 | 119
  Deterioration | 22 | 13

17. Secondary Outcome: Change From Baseline in PPBC at Week 12
Description: as for outcome 16
Time Frame: Baseline and Week 12
Population: FAS; N=participants with evaluable data; LOCF method was used for the statistical analyses of the FAS (change from baseline to Week 12).
Measure: Number; unit: Participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 368 | 360
Participants
  Improvement | 204 | 256
  No Change | 164 | 104
  Deterioration | 33 | 17
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Logistic regression determined the odds of improvement versus no improvement in PPBC score, where improvement was defined as a negative change from baseline; Covariates were treatment, study center, dosing time, age category, and baseline PPBC category; Odds Ratio (OR) = 2.506, 95% CI 2-sided [1.767 to 3.556]

18. Secondary Outcome: Change From Baseline in PPBC at Week 24
Description: as for outcome 16
Time Frame: Baseline and Week 24
Population: Not analyzed
Measure: Number; unit: Participants
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change From Baseline Patient Perception of Urgency Scale (PPUS) at Week 4
Description: PPUS: self-administered, single-item, questionnaire that measured the participant's perception of urinary urgency. It was sensitive to changes in perceptions of urinary urgency over time. Scale of 0 (usually not able to hold urine), 1 (usually able to hold urine [without leaking] until reaching toilet if go to toilet immediately), or 2 (usually able to finish what he/she was doing before going to toilet [without leaking]). Change = observation minus baseline. Improvement in PPUS defined as increase of 1 or more points in difference of scores relative to baseline.
Time Frame: Baseline and Weeks 4
Population: FAS; N=participants with evaluable data
Measure: Number; unit: Participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 370 | 361
Participants
  Improvement | 74 | 90
  No Change | 263 | 250
  Deterioration | 33 | 21

20. Secondary Outcome: Change From Baseline in PPUS at Week 8
Description: as for outcome 19
Time Frame: Baseline and Week 8
Population: FAS; N=participants with evaluable data
Measure: Number; unit: Participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 351 | 330
Participants
  Improvement | 95 | 111
  No Change | 224 | 194
  Deterioration | 32 | 25

21. Secondary Outcome: Change From Baseline in PPUS at Week 12
Description: as for outcome 19
Time Frame: Baseline and Week 12
Population: as for outcome 17
Measure: Number; unit: Participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 367 | 361
Participants
  Improvement | 109 | 133
  No Change | 226 | 200
  Deterioration | 32 | 28
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; LOCF; Test type: Superiority or Other; p = 0.0009, Regression, Logistic — Logistic regression determined the odds of improvement versus no improvement in PPBC score, where improvement was defined as an increase of 1 or more points in difference of scores relative to baseline; Covariates were treatment, study center, dosing time, age category, and baseline PPUS category; Odds Ratio (OR) = 1.916, 95% CI 2-sided [1.305 to 2.811]

22. Secondary Outcome: Change From Baseline in PPUS at Week 24
Description: as for outcome 19
Time Frame: Baseline and Week 24
Population: Not analyzed
Measure: Number; unit: Participants
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change From Baseline in Overactive Bladder Satisfaction Questionnaire (OAB-q) Symptom/Bother Score at Weeks 4, 8, 12, and 24
Description: OAB-q: self-administered, 33-item, questionnaire assessed how much participant was bothered by selected bladder symptoms during previous week. Each item rated by participant on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Raw scores transformed to a score from 0-100 where higher scores represented less favorable outcome. Change = baseline minus observation and higher scores were an improvement.
Time Frame: Baseline and Weeks 4, 8, 12, and 24
Population: FAS; N=participants with evaluable data; n=participants with evaluable data at specific time point. LOCF method was used for the statistical analyses of the FAS (change from baseline to Week 12). Change from baseline to Week 24 not analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 373 | 382
Scores on a scale
  Baseline (n=381, 373) | 52.90 (18.75) | 50.58 (19.35)
  Change at Week 4 (n=369, 358) | -9.03 (17.74) | -14.05 (18.37)
  Change at Week 8 (n=349, 328) | -12.86 (18.95) | -18.03 (19.25)
  Change at Week 12 (n=366, 357) | -12.16 (20.19) | -18.37 (21.38)
  Change at Week 24 | NA (NA) — Not Applicable (NA); Week 24 data collected change from baseline not calculated | NA (NA) — Week 24 data collected change from baseline not calculated
Statistical Analysis 1: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline symptom/bother score; Mean Difference (Final Values) = -7.12, 95% CI 2-sided [-9.65 to -4.59], Standard Error of Mean 1.29

24. Secondary Outcome: Change From Baseline in Overactive Bladder Satisfaction Questionnaire (OAB-q) Total Score at Weeks 4, 8, 12, and 24
Description: OAB-q: self-administered, 33-item, questionnaire assessed how much participant was bothered by selected bladder symptoms during previous week. Each item rated by participant on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Raw scores transformed to a score from 0-100 where higher scores represented less favorable outcome. Change = observation minus baseline and higher scores were an improvement.
Time Frame: Baseline and Weeks 4, 8, 12, and 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 373 | 379
Scores on a scale
  Baseline (n=373, 379) | 62.45 (20.20) | 64.42 (19.82)
  Change at Week 4 (n=367, 354) | 7.28 (15.48) | 10.24 (14.92)
  Change at Week 8 (n=348, 328) | 9.36 (17.98) | 12.96 (16.76)
  Change at Week 12 (n=363, 357) | 9.56 (18.75) | 13.19 (17.49)
  Change at Week 24 | NA (NA) — Change from Week 12 to Week 24 calculated instead of change from baseline to Week 24 | NA (NA) — Change from Week 12 to Week 24 calculated instead of change from baseline to Week 24
Statistical Analysis 1: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; Week 12 LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total health-related quality of life (HRQL) score; Mean Difference (Final Values) = 4.48, 95% CI 2-sided [2.24 to 6.73], Standard Error of Mean 1.14

25. Secondary Outcome: Change From Baseline in OAB-q Subscale Scores at Weeks 4, 8, 12, and 24
Description: OAB-q: self-administered, 33-item, questionnaire assessed how much participant bothered by bladder symptoms during previous week. Each item rated by participant on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Raw scores transformed to 0-100 score where higher scores were less favorable outcome. Questions 1-8 constituted symptom severity/bother score. Questions 9-33 constitute HRQL component, which included domains of coping, concern, sleep, and social function. Change = observation minus baseline and higher scores were an improvement.
Time Frame: Baseline and Weeks 4, 8, 12, and 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 380 | 374
Scores on a scale
  Coping at Baseline (n=380, 374) | 57.52 (24.36) | 58.31 (24.05)
  Coping Change at Week 4 (n=368, 358) | 8.35 (19.28) | 11.90 (17.98)
  Coping Change at Week 8 (n=348, 329) | 10.46 (20.96) | 14.98 (20.48)
  Coping Change at Week 12 (n=365, 358) | 10.60 (22.78) | 15.65 (21.52)
  Coping Change at Week 24 | NA (NA) — Week 24 data collected, change from baseline not analyzed. | NA (NA) — Week 24 data collected, change from baseline not analyzed.
  Concern at Baseline (n=380, 374) | 62.10 (23.32) | 64.67 (22.47)
  Concern Change at Week 4 (n=368, 358) | 7.96 (17.80) | 11.88 (18.20)
  Concern Change at Week 8 (n=348, 329) | 10.88 (21.23) | 15.39 (19.77)
  Concern Change at Week 12 (n=365, 358) | 11.25 (21.39) | 15.48 (20.23)
  Concern Change at Week 24 | NA (NA) — Week 24 data collected, change from baseline not analyzed. | NA (NA) — Week 24 data collected, change from baseline not analyzed.
  Sleep at Baseline (n=380, 374) | 53.79 (23.69) | 57.52 (23.83)
  Sleep Change at Week 4 (n=368, 358) | 7.31 (20.13) | 9.07 (18.61)
  Sleep Change at Week 8 (n=348, 329) | 9.01 (21.42) | 10.87 (20.07)
  Sleep Change at Week 12 (n=365, 358) | 9.36 (22.08) | 11.99 (21.33)
  Sleep Change at Week 24 | NA (NA) — Week 24 data collected, change from baseline not analyzed. | NA (NA) — Week 24 data collected, change from baseline not analyzed.
  Social at Baseline (n=380, 374) | 79.10 (21.84) | 81.02 (20.43)
  Social Change at Week 4 (n=368, 355) | 4.41 (16.01) | 6.25 (14.27)
  Social Change at Week 8 (n=349, 328) | 5.84 (18.58) | 8.17 (17.24)
  Social Change at Week 12 (n=364, 357) | 5.29 (18.56) | 7.02 (17.40)
  Social Change at Week 24 | NA (NA) — Week 24 data collected, change from baseline not analyzed. | NA (NA) — Week 24 data collected, change from baseline not analyzed.
Statistical Analysis 1: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; Coping Subscale at Week 12; LOCF; Test type: Superiority or Other; p = 0.0002, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline HRQL subscale score; Mean Difference (Final Values) = 5.39, 95% CI 2-sided [2.57 to 8.22], Standard Error of Mean 1.44
Statistical Analysis 2: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; Concern Subscale at Week 12; LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline HRQL subscale score; Mean Difference (Final Values) = 5.39, 95% CI 2-sided [2.84 to 7.93], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; Sleep Subscale at Week 12; LOCF; Test type: Superiority or Other; p = 0.0032, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline HRQL subscale score; Mean Difference (Final Values) = 4.09, 95% CI 2-sided [1.38 to 6.81], Standard Error of Mean 1.38
Statistical Analysis 4: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; Social Subscale at Week 12; LOCF; Test type: Superiority or Other; p = 0.0152, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline HRQL subscale score; Mean Difference (Final Values) = 2.51, 95% CI 2-sided [0.49 to 4.53], Standard Error of Mean 1.03

26. Secondary Outcome: Change From Week 12 in Overactive Bladder Satisfaction (OAB-S) Scale for Satisfaction With OAB Control at Week 24
Description: OAB-S: validated self-administered instrument that evaluated OAB medication expectations, daily life with OAB, and satisfaction with OAB medication and included 3 stand-alone items that assessed overall expectation, satisfaction, and willingness to continue treatment. Satisfaction coded on scale of 1-5: (1-very satisfied to 5-very dissatisfied). Coding reversed algorithmically and results transformed: total score range 0-100. Higher final response value associated with better satisfaction. Change = score at Week 24 minus score at Week 12 where higher scores indicated better satisfaction.
Time Frame: Weeks 12 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Fesoterodine/Fesoterodine: Participants received 12 weeks of fesoterodine 4 mg once daily (double-blinded), followed by 12 weeks of fesoterodine 4 mg once daily (open-label). During study, participants permitted 1 dose increase to 8 mg once daily (and 1 decrease from 8 mg back to 4 mg, if necessary).
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 330 | 301
Scores on a scale
  Week 12 | 44.97 (28.42) | 63.01 (24.16)
  Change at Week 24 | 21.22 (28.47) | 3.58 (20.27)
Statistical Analysis 1: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; LOCF; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Analysis determined the odds of responding on the OAB-S scale (satisfaction with OAB control) for Fesoterodine versus placebo, where a responder was defined as a response of 'satisfied' or better on all 7 questions at week 12; Covariates were treatment, study center, dosing time and age category; Odds Ratio (OR) = 3.537, 95% CI 2-sided [2.281 to 5.484]

27. Secondary Outcome: Change From Week 12 in OAB-S Scale for OAB Medication Expectation at Week 24
Description: OAB-S: evaluated OAB medication expectations, daily life with OAB, and satisfaction with OAB medication. Included 3 stand-alone items that assessed overall expectation, satisfaction, and willingness to continue treatment. Medication expectation coded on scale 1=Greatly exceeds my expectations to 5=Does not meet my expectations at all. Coding reversed by subtracting initial response value from 6, so higher final response value associated with better fulfilment of OAB medication expectations.
Time Frame: Weeks 12 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 330 | 301
Scores on a scale
  Week 12 | 2.21 (1.07) | 2.85 (1.10)
  Change at Week 24 | 0.74 (1.22) | 0.17 (1.04)
Statistical Analysis 1: Comparison: Placebo/Fesoterodine vs Fesoterodine/Fesoterodine; LOCF; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Analysis determined the odds of responding on the OAB-S scale (OAB medication expectation) for Fesoterodine versus placebo, where a responder was defined as a response of 'satisfied' or better on all 7 questions at week 12; Covariates were treatment, study center, dosing time and age category; Odds Ratio (OR) = 2.881, 95% CI 2-sided [2.045 to 4.058]

28. Secondary Outcome: Change From Baseline in King's Health Questionnaire (KHQ) Domain Scores at Week 12
Description: KHQ: self-administered questionnaire contained 21 questions scored in 9 domains (general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy, severity of urinary symptoms). Range: 0-100, where 0=best outcome/response and 100=worst outcome/response. Change = observation minus baseline, where lower scores indicated better outcome/response.
Time Frame: Baseline and Week 12
Population: FAS; N=participants with evaluable data at sites in the United Kingdom only; n=participants with evaluable data for specific KHQ category. LOCF method used for statistical analyses of the FAS (change from baseline to Week 12).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 23 | 32
Scores on a scale
  Baseline General Health Perception (n=23, 32) | 35.87 (19.69) | 25.00 (17.96)
  Change at Week 12 General Hlth Perception n=21, 29 | -2.38 (15.62) | 2.59 (13.93)
  Baseline Incontinence Impact (n=23, 32) | 75.36 (25.06) | 73.96 (29.00)
  Change at Week 12 Incontinence Impact (n=21, 29) | -12.70 (32.45) | -16.09 (34.06)
  Baseline Role Limitations (n=22, 32) | 48.48 (34.85) | 46.35 (30.15)
  Change at Week 12 Role Limitations (n=20, 29) | -10.83 (45.33) | -12.64 (25.45)
  Baseline Physical Limitations (n=22, 32) | 50.76 (31.49) | 44.79 (32.91)
  Change at Week 12 Physical Limitations (n=20, 29) | -13.33 (30.40) | -13.79 (28.20)
  Baseline Social Limitations (n=22, 32) | 24.75 (23.43) | 29.86 (33.89)
  Change at Week 12 Social Limitations (n=20, 29) | -7.50 (23.17) | -8.62 (24.20)
  Baseline Personal Relationships (n=16,17) | 15.63 (28.85) | 19.61 (27.15)
  Change at Week 12 Personal Relationship (n=11, 14) | 4.55 (18.40) | -5.95 (18.03)
  Baseline Emotions (n=22, 32) | 32.32 (25.64) | 32.64 (29.18)
  Change at Week 12 Emotions (n=20, 29) | -2.78 (28.58) | -6.51 (25.63)
  Baseline Sleep/Energy (n=22, 32) | 46.97 (27.04) | 57.29 (27.74)
  Change at Week 12 Sleep/Energy (n=20, 29) | -8.33 (26.21) | -11.49 (23.61)
  Baseline Severity USS (n=22, 32) | 43.94 (22.69) | 44.38 (25.99)
  Change at Week 12 Severity USS (n=20, 29) | -2.00 (18.99) | -8.51 (16.70)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; General Health Perception; LOCF; Test type: Superiority or Other; p = 0.3163, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = 4.18, 95% CI 2-sided [-4.13 to 12.49], Standard Error of Mean 4.12
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Incontinence Impact; LOCF; Test type: Superiority or Other; p = 0.4698, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = -6.29, 95% CI 2-sided [-23.70 to 11.11], Standard Error of Mean 8.63
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Role Limitations; LOCF; Test type: Superiority or Other; p = 0.5321, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = -5.85, 95% CI 2-sided [-24.58 to 12.88], Standard Error of Mean 9.28
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Physical Limitations; LOCF; Test type: Superiority or Other; p = 0.6523, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = -3.81, 95% CI 2-sided [-20.74 to 13.12], Standard Error of Mean 8.39
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Social Limitations; LOCF; Test type: Superiority or Other; p = 0.6344, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = 3.26, 95% CI 2-sided [-10.47 to 16.99], Standard Error of Mean 6.80
Statistical Analysis 6: Comparison: Placebo vs Fesoterodine; Personal Relationships; LOCF; Test type: Superiority or Other; p = 0.2013, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = -11.11, 95% CI 2-sided [-28.71 to 6.49], Standard Error of Mean 8.38
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Emotions; LOCF; Test type: Superiority or Other; p = 0.3831, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = -6.07, 95% CI 2-sided [-19.96 to 7.83], Standard Error of Mean 6.88
Statistical Analysis 8: Comparison: Placebo vs Fesoterodine; Sleep/Energy; LOCF; Test type: Superiority or Other; p = 0.5167, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = 4.46, 95% CI 2-sided [-9.30 to 18.23], Standard Error of Mean 6.82
Statistical Analysis 9: Comparison: Placebo vs Fesoterodine; Severity of Urinary Symptoms; LOCF; Test type: Superiority or Other; p = 0.0532, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline total domain score; Mean Difference (Final Values) = -10.19, 95% CI 2-sided [-20.53 to 0.15], Standard Error of Mean 5.12

29. Secondary Outcome: Change From Baseline in EQ-5D- Health State Profile Utility Score at Week 12
Description: EQ-5D: participant rated questionnaire to assess HRQL in terms of single index value. Visual Analogue Scale (VAS) component rated current health state on scale from 0 (worst imaginable health state) to 100 (best imaginable health state). For each question, scores categorized into 3 levels of response, level 1=no health problems, 2=some problems and 3= extreme problems, and health state profile utility score derived from these, which could range from 1 prefect health to -0.594 worst possible health. Change = observation minus baseline, where higher scores indicated a better health state.
Time Frame: Baseline and Week 12
Population: FAS; N=participants with evaluable data; n=participants with evaluable data a specified time point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 381 | 373
Scores on a scale
  Baseline (n=381, 373) | 0.7825 (0.2246) | 0.8092 (0.2068)
  Change at Week 12 (n=362, 346) | 0.0230 (0.1963) | 0.0064 (0.1854)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Test type: Superiority or Other; p = 0.8959, ANCOVA; Covariates were treatment, study center, dosing time, age category, and baseline single utility score; Mean Difference (Final Values) = 0.0016, 95% CI 2-sided [-0.0229 to 0.0262], Standard Error of Mean 0.0125

30. Secondary Outcome: Change From Baseline in EQ-5D- Each Dimension Score at Week 12
Description: EQ-5D: participant rated questionnaire to assess HRQL in terms of a single utility score. Health State Profile component assessed level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicated better health state; 3 indicated worst health state. Scoring formula assigned utility value for each domain in profile. Score was transformed and results in total score could have ranged from -0.594 to 1.000; Change = observation minus baseline, where higher scores indicated a better health state.
Time Frame: Baseline and Week 12
Population: Not analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) at Week 12
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranged from 0 - 30, higher score indicated better cognitive state. Change = observation minus baseline where higher scores indicated better cognitive functioning.
Time Frame: Baseline and Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 382 | 374
Scores on a scale
  Baseline | 28.09 (1.98) | 28.20 (1.94)
  Change at Week 12 | 0.23 (1.82) | 0.24 (1.76)

32. Other Pre Specified Outcome: Percentage of Participants With Improvement at Week 24
Description: Patient Treatment Benefit Scale (PTBS): single-item scale assessed fesoterodine efficacy and safety in participants with overactive bladder. Participants asked to compare their present condition with their condition before start of trial: "My condition has been: 1=Greatly Improved; 2=Improved; 3=Not Changed; 4=Worsened, During Treatment." Treatment Response was set to "Yes" if the first 2 categories (1 or 2) of the scale selected and "No" if the last 2 categories (3 or 4) were selected. Improvement was defined as a rating of 1 or 2.
Time Frame: Pre-baseline and Week 24
Population: Not analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 0 | 0

33. Other Pre Specified Outcome: Change From Baseline in Number of Micturition-Related Urgency Episodes Per 24 Hours at Week 24
Description: Number of micturition-related urgency episodes per 24 hours calculated as number of micturitions with USS rating of >=3 divided by number of days that diary data was collected at that visit. USS rating of 3: Moderate feeling of urgency, 4: Severe feeling of urgency, 5: Unable to hold; leak urine). Change = observation minus baseline, where lower scores were an improvement/decrease in micturition-related urgency episodes.
Time Frame: Baseline and Week 24
Population: FAS; N=participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 332 | 305
Episodes per 24 hours | -4.24 (4.62) | -4.07 (4.23)

34. Other Pre Specified Outcome: Change From Baseline in Mean Number of Severe Micturition-Related Urgency Episodes Per 24 Hours at Week 24
Description: Severe micturition-related urgency episodes defined as those with the USS rating >=4. USS rating of 4: Severe feeling of urgency and 5: Unable to hold; leak urine. Change = observation minus baseline, where lower scores were an improvement/decrease in micturition-related urgency episodes.
Time Frame: Baseline and Week 24
Population: FAS; N=participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 332 | 305
Episodes per 24 hours | -2.57 (4.37) | -2.41 (3.30)

35. Other Pre Specified Outcome: Change From Baseline in Number of Nocturnal Micturitions Per 24 Hours at Week 24
Description: Nocturnal micturitions were defined as micturitions with USS rating 1-5 that occurred between the time the participant went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. Calculated as number of nocturnal micturitions divided by number of diary days collected at that visit. Change = observation minus baseline, where lower scores were an improvement/decrease in nocturnal micturitions.
Time Frame: Baseline and Week 24
Population: FAS; N=participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Micturitions per 24 hours
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 332 | 305
Micturitions per 24 hours | -0.60 (1.24) | -0.67 (1.18)

36. Other Pre Specified Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 24
Description: Micturitions include episodes of voluntary micturition and episodes of UUI. UUI episodes defined as those micturitions with USS rating of 5 (unable to hold; leak urine) in the diary in participants with UUI at baseline. Change = observation minus baseline, where lower scores were an improvement/decrease in micturitions.
Time Frame: Baseline and Week 24
Population: FAS; N=participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Micturitions per 24 hours
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 333 | 305
Micturitions per 24 hours | -2.28 (2.89) | -2.36 (2.57)

37. Other Pre Specified Outcome: Change From Baseline in Mean Number of UUI Episodes Per 24 Hours at Week 24
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: FAS; N=participants with evaluable data.
Measure: Median (Full Range); unit: Episodes per 24 hours
Arm/Group | Placebo/Fesoterodine | Fesoterodine/Fesoterodine
Number analyzed (Participants) | 333 | 305
Episodes per 24 hours | 0.0 [-26.7 to 13.7] | 0.0 [-14.3 to 4.0]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 subject and as nonserious in another subject, or 1 subject may have experienced both a serious and nonserious event during the study.
Groups:
- Placebo Double-Blind: Participants received matched placebo once daily from baseline to Week 12 (double-blinded)
- Fesoterodine Double-Blind: Participants received fesoterodine 4 mg once daily from baseline to Week 12 (double-blinded)
- Festerodine/Fesoterodine Open-Label: Participants received 12 weeks of fesoterodine 4 mg once daily (double-blinded), followed by 12 weeks of fesoterodine 4 mg once daily (open-label). Serious adverse events (SAEs) and non-serious adverse events (AEs) reported reported for these participants only during the open-label phase.
- Placebo/Fesoterodine Open-label: Participants received 12 weeks of matched placebo (double-blinded), followed by 12 weeks of fesoterodine 4 mg once daily (open-label). SAEs and non-serious AEs reported for these participants only during the open-label phase.
Arm/Group | Placebo Double-Blind | Fesoterodine Double-Blind | Festerodine/Fesoterodine Open-Label | Placebo/Fesoterodine Open-label
Serious Adverse Events (participants affected / at risk) | 9/393 | 14/392 | 11/313 | 7/341
Other Adverse Events (participants affected / at risk) | 71/393 | 187/392 | 49/313 | 119/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Double-Blind (N=393) | Fesoterodine Double-Blind (N=392) | Festerodine/Fesoterodine Open-Label (N=313) | Placebo/Fesoterodine Open-label (N=341)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Optic nerve infarction (Eye disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral polyp (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Aneurysm ruptured (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Double-Blind (N=393) | Fesoterodine Double-Blind (N=392) | Festerodine/Fesoterodine Open-Label (N=313) | Placebo/Fesoterodine Open-label (N=341)
Constipation (Gastrointestinal disorders) | 10 | 35 | 5 | 21
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 21 | 133 | 21 | 95
Dyspepsia (Gastrointestinal disorders) | 2 | 9 | 3 | 4
Nausea (Gastrointestinal disorders) | 4 | 9 | 2 | 1
Fatigue (General disorders) | 10 | 9 | 0 | 4
Nasopharyngitis (Infections and infestations) | 9 | 12 | 6 | 2
Urinary tract infection (Infections and infestations) | 7 | 10 | 14 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 2 | 4 | 3
Dizziness (Nervous system disorders) | 4 | 14 | 2 | 6
Headache (Nervous system disorders) | 5 | 11 | 0 | 7
Hypertension (Vascular disorders) | 8 | 7 | 2 | 7

LIMITATIONS AND CAVEATS:
The descriptive statistics and analyses of outcome measure 12 as defined in the protocol are not presented. Results are presented as defined in the statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.